CLINICAL TRIAL: NCT05525377
Title: Better Living With Non-memory-led Dementia: Feasibility Study on the Effects of a Blended Online Training Course for Carers of People With Atypical AD and FTD.
Brief Title: Better Living With Non-memory-led Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RDSImpact_ws4feasibility
Record Dates: First submitted 2022-08-12; First posted 2022-09-01 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2022-08

CONDITIONS: Primary Progressive Aphasia; Frontotemporal Dementia; Alzheimer Disease
Keywords: "Posterior Cortical Atrophy"
MeSH Terms: conditions — Aphasia, Primary Progressive; Frontotemporal Dementia; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Subjects in the intervention group receive access to an online training and educational phenotype-specific programme on how to support their relative with non-memory-led dementia. The online course consists on 6 modules to complete in 7 weeks. A course facilitator is available throughout the duration of the intervention to support participants.
  Interventions: Behavioral: Better living with non-memory led dementia course
- Treatment as usual (TAU) (No Intervention): The "treatment as usual" group does not receive access to the educational programme.

INTERVENTIONS:
Behavioral: Better living with non-memory led dementia course — Caregivers online training and educational phenotype-specific programme on how to support people with non-memory-led dementia.
  Arms: Intervention

SUMMARY:
This is a feasibility study on the effects of an online-based training and education programme for carers of people with posterior cortical atrophy (PCA), primary progressive aphasia (PPA) and behavioural-variant frontotemporal dementia (bvFTD).

DETAILED DESCRIPTION:
The purpose of this study is:

To evaluate the feasibility of an online training course for carers of people with PCA, PPA, and bvFTD. Feasibility measures will focus on the recruitment process and measurement tools.

To determine the acceptability of an online training course for carers of people with PCA, PPA and bvFTD.

The study will involve 6 online modules over the course of 7 weeks. All sessions will take place over the internet, using an online platform. A research team member (facilitator) will be available to assist participants over the course completion.

ELIGIBILITY:
Inclusion Criteria:

1. . Adults (18+) who self-identify as an unpaid carer (partners, children, friends, etc.) of someone with PPA, PCA or bvFTD who is not living in a full-time care facility.
2. . The care recipient has to have a confirmed diagnosis of dementia (through self-report of the carer, to reflect the 'real world' application of the intervention).

Exclusion Criteria:

1. . Those unable to comprehend written English
2. . Those with no access to the internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Study feasibility | Since June 2022 to January 2023 (8 months)
  Feasibility of recruitment process and measurement tools (e.g., number of people agreeing to be sent information about the study, time taken to fill in questionnaires).
Acceptability | Since June 2022 to January 2023 (8 months)
  Prospective and retrospective acceptability (e.g., reasons for not taking part, task completion rate after every module)

SECONDARY OUTCOMES:
WHO 5 Wellbeing Index | Change from baseline to 8 weeks and 3 months
  Short self-reported measure of current mental wellbeing (ranging from 0 (minimun) to 25 (maximun) scores). 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Generalized Anxiety Disorder scale (GAD-7) | Change from baseline to 8 weeks and 3 months
  Generalized Anxiety Disorder scale (ranging from 0 (minimun) to 21 (maximun) scores). Higher scores indicates higher anxiety.
Patient Health Questionnaire (PHQ-9) | Change from baseline to 8 weeks and 3 months
  Assesses depression severity (ranging from 0 (minimun) to 27 (maximun) scores. Higher scores indicate higher depression.
De Jong Gierveld Loneliness Scale | Change from baseline to 8 weeks and 3 months
  Measure variations in total loneliness score ranging from 0 (minimun) to 11 (maximun) scores. 0 meaning not lonely and 100 very severe lonely score.
Lubben Social Network Scale | Change from baseline to 8 weeks and 3 months
  Brief instrument designed to gauge social isolation in older adults by measuring perceived social support received by family and friends. Ranging from 0 (minimun) to 60 (maximun) scores. Higher scores represent higher social network.
Pearling Mastery Scale | Change from baseline to 8 weeks and 3 months
  Measures the extent to which an individual regards their life chances as being under their personal control. Ranging from 7 (minimun) to 28 (maximun) scores. Higher scores indicate greater levels of mastery.
Caregiver self-efficacy scale | Change from baseline to 8 weeks and 3 months
  Measures caregivers' beliefs about their ability to carry out behaviors such as obtaining respite, responding to disruptive patient behaviors, etc. Ranging from 0 (minimun) to 100 (maximun) scores. Higher scores reflect higher confidence.
Dementia Management Strategies Scale | Change from baseline to 8 weeks and 3 months
  Instrument to appraise 3 care styles of caregivers: 1) Active management, 2) Criticism and 3) Encouragement. Ranging from 34 (minimun) to 170 (maximun). Higher scores mean a greater presence of behaviours associated to the the corresponding caregiver style.
The quality of carer-partner relationship scale | Change from baseline to 8 weeks and 3 months
  Scale that measures closeness in a relationship. Ranging from 14 (minimun) to 70 (maximun). Higher scores reflect higher quality of carer-partner relationship.
Questions about perceived burden and ethicality | At 8 weeks post-randomisation and 3 month follow up
  Tailored questions administered in a purposed-built interview. They
Health economics questions | At 8 weeks post-randomisation and 3 month follow up
  Tailored questions administered in a purposed-built interview.

CONTACTS AND LOCATIONS:
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suarez-Gonzalez A, John A, Brotherhood E, Camic PM, McKee-Jackson R, Melville M, Sullivan MP, Tudor-Edwards R, Windle G, Crutch S, Hoare Z, Stott J; Rare Dementia Support Impact team. "Better Living with Non-memory-led Dementia": protocol for a feasibility randomised controlled trial of a web-based caregiver educational programme. Pilot Feasibility Stud. 2023 Oct 11;9(1):172. doi: 10.1186/s40814-023-01403-1. PMID 37821924